CLINICAL TRIAL: NCT00924963
Title: Comparison of J-Tip® Jet Injection of 1% Buffered Lidocaine, 4% Lidocaine Topical Cream, and J-Tip® Jet Injection of Placebo Prior to Venipuncture and Peripheral Intravenous Catheter Insertion in a Pediatric Emergency Department
Brief Title: J-Tip® Jet Injection of 1% Buffered Lidocaine or Saline Versus 4% Lidocaine Cream Before Venipuncture or IV Insertion
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study ended due to lack of funding.
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2008-0922
Record Dates: First submitted 2009-06-18; First posted 2009-06-19 (Estimated); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Pain
Keywords: Pain of venipuncture or IV insertion
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Jet injection lidocaine (Experimental): J-Tip jet injection of 1% buffered lidocaine
  Interventions: Device: J-Tip jet injector
- Jet injection saline (Placebo Comparator): J-Tip jet injection of sterile saline
  Interventions: Device: Jet injection saline
- Lidocaine cream (Active Comparator): Lidocaine 4%cream applied for 30 minutes prior to IV insertion or venipuncture
  Interventions: Drug: lidocaine cream

INTERVENTIONS:
Device: J-Tip jet injector — 0.2ml 1%buffered lidocaine delivered by jet injector
  Other Names: J-Tip jet injector with 1% buffered lidocaine
  Arms: Jet injection lidocaine
Device: Jet injection saline — 0.2ml saline delivered via J-Tip jet injection
  Other Names: J-Tip Jet injection with saline
  Arms: Jet injection saline
Drug: lidocaine cream — 4% lidocaine cream applied for 30 minutes to the skin
  Other Names: 4% lidocaine cream
  Arms: Lidocaine cream

SUMMARY:
To measure and compare pain associated with venipuncture and peripheral intravenous catheter insertion among pediatric emergency department patients randomized to treatment with one of three different pain-reduction strategies: J-Tip® jet injection of 1% buffered lidocaine, J-Tip® jet injection of sterile saline, or application of 4% lidocaine topical cream. The investigators hypothesize that J-Tip® jet injection of 1% buffered lidocaine will provide superior local anesthesia compared to saline or lidocaine cream.

DETAILED DESCRIPTION:
Background: Venipuncture and PIVC insertion are the most common procedures performed in the pediatric emergency department. They are painful procedures, and frequently no local anesthesia is provided. The American Academy of Pediatrics Committee on Pediatric Emergency Medicine and Section on Anesthesiology and Pain Medicine has recommended that local anesthesia be provided, but a variety of barriers exist which have prevented implementation of this recommendation.

Specific Aims: To measure and compare pain associated with venipuncture and peripheral intravenous catheter insertion among pediatric emergency department patients randomized to treatment with one of three different pain-reduction strategies: J-Tip® jet injection of 1% buffered lidocaine, J-Tip® jet injection of sterile saline, or application of 4% lidocaine topical cream.

Methods: This study is a partially blinded, placebo controlled, randomized controlled clinical trial in the pediatric emergency department. The comparison of J-Tip® jet injection of 1% buffered lidocaine to J-Tip® jet injection of sterile saline is double blinded, while the comparison of jet injection to 4% lidocaine topical cream is not blinded. Forty-four patients per group will be enrolled, and a VAS self-reported measurement will be recorded for the pain of venipuncture or PIVC insertion following the appropriate treatment. As well, success of the procedure and complications of treatment will be recorded.

Results: Pain scores will be analyzed by pairwise comparisons using a t-test and pooled comparisons using ANOVA. Demographics will be assessed to determine baseline differences among the three groups. Chi square and regression analysis will be performed on demographic differences to determine significance if necessary. Final pain results will be reported as mean, standard deviation, and p-value. Demographics will be reported as number, percent of patients, and p-value (if a difference exists).

ELIGIBILITY:
Inclusion Criteria:

* Children aged seven to twenty-one years old requiring venipuncture or PIVC insertion as part of their emergency department care are eligible for the study.

Exclusion Criteria:

* Lidocaine allergy,
* TegadermTM allergy,
* Glasgow Coma Score (GCS) less than 15,
* Pain at the proposed site for the procedure,
* Requirement of a PIVC or venipuncture immediately due to illness acuity,
* Inability to complete a self-reported pain scale (VAS, visual analogue scale),
* Patients who do not speak and understand English, OR
* Previous enrollment in the study.

Ages: 7 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Jet injection of 1% buffered lidocaine to 4% lidocaine topical cream to measure the effectiveness of jet injection of lidocaine as a local anesthetic prior to venipuncture and PIVC insertion | 30 minutes
  1. Pain associated with venipuncture or PIVC insertion after pre-treatment with jet injection of 1% buffered lidocaine versus 4% lidocaine topical cream

SECONDARY OUTCOMES:
Jet injection of 1% buffered lidocaine to jet injection of saline to assess and measure a potential placebo effect not measured in prior studies | 30 minutes
  Pain associated with venipuncture or PIVC insertion after pre-treatment with jet injection of 1% buffered lidocaine versus jet injection of sterile saline
Second attempt pain scores (if occurred) among the three groups and between their first and second VAS scores | 30 minutes
  compare pain scores across groups if a second attempt was made using VAS scores
The success of venipuncture or PIVC insertion with all anesthetic techniques | 30 minutes
  Compare all types of anesthetics during venipuncture or PIVC
Variety of locations of successful venipuncture or PIVC insertion after jet injection use | 30 minutes
  compare successful venipunctures across locations
Measurement of complication rate after jet injection use | 1 hour
  Compare variability of complications that arise post injection across groups

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Spanos, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Srikant Iyer, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Liberty Township Emergency Department, Liberty Township, Ohio, United States